CLINICAL TRIAL: NCT00519623
Title: Pharmacokinetic/Pharmacodynamic Study of the PassPort(R) Transdermal Insulin Delivery System in Type 1 Diabetes Patients
Brief Title: Transdermal Basal Insulin Patch Study in Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altea Therapeutics (Industry)
Responsible Party: Alan Smith, Vice President, Product Development, Clinical R&D, and Project Management, Altea Therapeutics Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN2007001
Record Dates: First submitted 2007-08-02; First posted 2007-08-22 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; insulin; blood sugar; type 1 diabetes; insulin dependent diabetes; transdermal
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PassPort(R) Transdermal Insulin Delivery System (Experimental)
  Interventions: Other: PassPort(R) Transdermal Insulin Delivery System

INTERVENTIONS:
Other: PassPort(R) Transdermal Insulin Delivery System — The PassPort(R) Transdermal Insulin Delivery System is a drug-device combination product used to create micropores in the skin to enable transdermal delivery of insulin.

SUMMARY:
This study is designed to evaluate the pharmacokinetics/pharmacodynamics of an investigational basal insulin patch in type 1 diabetes patients.

DETAILED DESCRIPTION:
The study is looking for patients that meet the following criteria:

* Duration of type diabetes greater than or equal to 10 years
* HbA1C less than or equal to 9.0%
* C-peptide negative
* Ages 18 - 65, male or female
* Body Mass Index (BMI) 18.5 - 32
* Non-smoker
* No advanced diabetes complications
* Not pregnant or breast feeding

ELIGIBILITY:
Inclusion Criteria:

* Duration of type 1 diabetes greater than or equal to 10 years
* HbA1c less than or equal to 9.0%
* C-peptide negative
* Ages 18 - 65, male or female
* BMI 18.5 - 32
* Non- smoker
* No advance diabetes complications
* Not pregnant or breast feeding

Exclusion Criteria:

* Arm or leg rashes, open wounds, or skin conditions
* Psychiatric disorders
* Participation in a clinical research trial in last 3 months
* Clinically significant acute illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Spratlin, M.D., Principal Investigator — Altea Therapeutics
Locations (1):
- Altea Therapeutics Clinical Research Center, 387 Technology Circle, NW, Suite 100, Atlanta, Georgia, United States

REFERENCES:
- [Result] Smith, A, Zerkel, K, Roerig, P, Mills, S, Humphries, C, Durland, R, Spratlin, V, "Transdermal Delivery of Insulin in Patients with Type 1 Diabetes," American Diabetes Association 68th Scientific Sessions, Abstract 309-OR, Diabetes 57 Supplement 1:A88, 2008.
- See also: Altea website — http://www.alteatherapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for the IN2007001 study were recruited between August 2007 and November 2007 by the Phase 1 Clinical Research Unit.
Pre-assignment Details: Subjects stopped intermediate/long-acting insulin 48 hours prior to treatment or discontinued use of their insulin pump when they arrived for the treatment. There was a run-in period in which IV insulin lispro was administered to achieve a glucose clamp target of 100 mg/dL prior to application of the patch.
Groups:
- Transdermal Patch: PassPort(r) Transdermal Insulin Delivery System
Period: Overall Study
Arm/Group | Transdermal Patch
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Patch
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of the PassPort(R) Transdermal Insulin Delivery System in Type 1 Diabetes Patients (Cmax)
Description: Study IN2007001 is designed to evaluate the PK/PD of the PassPort(R) Transdermal Insulin Delivery System in type 1 diabetes patients. The PK was determined by analysis of serum insulin assay values. The mean Cmax was reported.
Time Frame: Samples were collected at -1,-0.25, 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 7.0, 8.0, 9.0, 10.0, 11.0, 12.0, 12.5, 13.0, 14.0, 15.0, 16.0 hours
Population: Number of subjects completed
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Transdermal Patch
Number analyzed (Participants) | 8
uU/mL | 33.0 (6.3)

2. Secondary Outcome: Skin Response to the Application of the PassPort(R) Transdermal Insulin Delivery System in Type 1 Diabetes Patients
Description: Skin response was evaulated by visual skin scoring using a modified Draize scale and transepidermal water loss (TEWL) measurements. The transdermal insulin patch was well-tolerated with mild transient erythema at the application site.
Time Frame: Time Points: prior to microporation, after microporation, after patch removal, 24 hours after patch removal, and 7 days after patch removal
Reporting Status: Not Posted, anticipated posting 2010-11
Measure: Mean (Standard Deviation); unit: TEWL (gH2O/m2/h)

3. Primary Outcome: Pharmacodynamics of the PassPort(R) Transdermal Insulin Delivery System in Type 1 Diabetes Patients (GIRmax)
Description: Study IN2007001 is designed to evaluate the PK/PD of the PassPort(R) Transdermal Insulin Delivery System in type 1 diabetes patients. The PD was determined by analysis of glucose infusion rates required to maintain the glucose clamp level of 100 mg/dL. The mean GIRmax was reported.
Time Frame: Glucose infusion rates were adjusted every 10 minutes as necessary
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Transdermal Patch
Number analyzed (Participants) | 8
mg/kg/min | 4.9 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study treatment until the last follow up visit (7 days after patch removal).
Description: Systematic assessments of adverse events were performed throughout the study via clinical staff assessments/questions and laboratory testing. In addition, adverse events were self-reported by subjects throughout the study.
Arm/Group | Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Patch (N=9)
Headache (Nervous system disorders) | 2 (3)
IV Site Pain/Swelling (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a small exploratory study to evaluate the PK, PD and tolerability of a selected Basal Insulin PassPort(r) System configuration in C-peptide negative type 1 diabetes subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is restricted from using, disclosing, presenting or publishing trial information without the prior written consent from the Sponsor.

PI is not an employee of the Sponsor but was paid to conduct the study at the Sponsor's Phase 1 Clinical Resarch Unit.